Official title: Capitalizing on the Strengths of Persons With Rheumatoid Arthritis to Improve Health and Wellness

Brief title: Feasibility of a Mobile Application to Support Reflection and Dialog About Strengths in People With Chronic Illness

NCT03437863

Date: 2021-03-19

## Study protocol and statistical analysis plan

Self-management of chronic illness can be highly demanding and people need to mobilize their personal strengths in order to live well with their condition. A mobile application was designed in collaboration with people with chronic illness and health care providers with the aims to support awareness of patients' strengths and patient-provider dialogues that include strengths. The aim of the present study is to evaluate with mixed methods the perceived usefulness and usability of the application and potential effects of the application on patients.

In this pre-post design pilot study participants will be recruited from self-management courses for people with rheumatic diseases. Before using the application participants will be asked to report their strengths in a written format. After using the mobile application to reflect on their strengths the participants will be interviewed about their experience of using the application and on the task of reflecting on their strengths. They will also be asked to fill out a questionnaire on perceived usefulness and user-friendliness. Before and after using the application the participants fill out questionnaires on emotions (Positive and Negative Affective Scale) and self-efficacy (The Arthritis Self-efficacy Scale). All interviews will be audio-taped and analyzed with a qualitative approach. Descriptive analysis will be applied for quantitative data.

## Note after study completion

The reason for the registration of this non-clinical study in the register is the original plan to include a clinical sub-study with healthcare provider-patient pairs using the application in clinical practice. Due to practical issues no participants were recruited in the clinical part of the project. The non-clinical feasibility pilot study (n=12) is published without referral to the clinical registration number since it was not considered a clinical study. The reference is:

Kristjansdottir, O. B., Børøsund, E., Westeng, M., Ruland, C., Stenberg, U., Zangi, H. A., ... & Mirkovic, J. (2020). Mobile App to Help People With Chronic Illness Reflect on Their Strengths: Formative Evaluation and Usability Testing. *JMIR formative research*, 4(3), e16831.

Date: 2021-03-19